CLINICAL TRIAL: NCT06853561
Title: Co-work Design: A Structural Approach to Reduce Individual Work Stress in Healthcare Professionals in Hospital Settings
Brief Title: Reducing Individual Work Stress in Healthcare Professionals Through Exchange of Job Resources
Status: Recruiting | Type: Observational
Sponsor: Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Luisa Solms, Postdoctoral researcher, Erasmus University Rotterdam
Other Study IDs: ETH2425-0324; 14160503.001 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2025-02-17; First posted 2025-03-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Job Crafting
Keywords: job crafting; work-related well-being; healthcare; nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study focuses on prosocial job crafting as a novel strategy to reduce burnout and foster well-being among nurse professionals. Specifically, we will examine whether prosocial job crafting enhances individual and team-level well-being by increasing own and others' resources.

DETAILED DESCRIPTION:
Below, we provide more information on the study design, study procedure, data collection, data management, and data analysis.

Study Design:

Type: Prospective, longitudinal, observational diary study. Duration: 10 workdays of daily surveys with a baseline survey at the start (Day 0).

Setting: Online survey tool (Castor), accessible via smartphones.

Study Procedure:

Day 0 - Baseline Survey: Collects demographic data and job-related information.

Days 1-10 - Daily Surveys:

Workday Verification: Confirmation of work on that day.

In addition to the outcomes listed under primary and secondary outcome measures, daily surveys will include measures of:

Prosocial Job Crafting: 12 items adapted to measure crafting behaviors to benefit other team members, using the Prosocial Job Crafting Measure (PSJCM).

Psychological Capital: 12 items measuring hope, self-efficacy, optimism, and resilience, using a shortened version of the Psychological Capital Questionnaire (PCQ).

Day 11 - Post-Study Survey: Summary of results and feedback opportunity.

Data Collection:

Survey Platform: Mobile-friendly (Castor). Questionnaire Format: Self-report measures adapted for daily context.

Data Management:

Anonymity: Participants are assigned anonymous codes for data matching. Confidentiality: Data is securely stored with access only for researchers on the project.

Statistical Analysis:

Multilevel modeling will be used to analyze the nested nature of daily data and relationships between job crafting, resource exchange, and work outcomes.

ELIGIBILITY:
Eligibility Criteria:

* Employees (nurse professionals) working in a team-based work environment (hospital setting).
* Participants must be able to complete daily surveys in the designated timeframe (end of each workday).

Exclusion Criteria:

* Part-time workers with small contracts (less than 3 days a week) or individuals not engaged in team-based work.
* Participants who do not complete the baseline survey or a minimum of 5 daily surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurse professionals working in an EU hospital.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Burnout | From the start of the study (i.e., at baseline, day 0) to the end of the study (i.e., at day 10).
  Burnout symptoms will be assessed using the ultra-short version of the Burnout Assessment Tool (BAT4) consisting of 4 items. The tool assesses perceptions of symptoms like exhaustion, mental distance, emotional impairment, and cognitive impairment based on self-reported responses. Notably, the different symptoms (e.g., exhaustion) are combined into a composite score to give an overall burnout measure rather than being treated as separate outcomes.
Work engagement | From start of study (i.e., at baseline, day 0) to end of study (i.e., at day 10).
  Work engagement will be assessed using a shortened, 3-item version of the Utrecht Work Engagement Scale (UWES), which captures a work-related and positive state of mind, characterized by vigor, dedication, and absorption. Items will be combined into a composite score to give an overall work engagement measure.
Flourishing | From the start of the study (i.e., at baseline, day 0) to the end of the study (day 10).
  Flourishing will be assessed with Diener's 8-item Flourishing Scale. The scale captures self-perceived success in important areas of life, such as relationships, self-esteem, purpose, and optimism. The score for flourishing is calculated by averaging the responses to these 8 items, with higher scores reflecting greater flourishing.
Job Resources Exchange | From the start of the study (i.e., at baseline, day 0) to the end of the study (day 10).
  Frequency of job resources exchange with other team members will be assessed based on scale developed by Edelmann and colleagues (not published). The scale assesses the extent to which individuals provide and receive feedback and knowledge to and from other members of their team.

SECONDARY OUTCOMES:
Workload | From the start of the study (i.e., at baseline, day 0) to end of the study (i.e., day 10).
  Workload will be measured with five items from the Questionnaire on the Experience and Evaluation of Work (QEEW). Responses will be combined into a composite score.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data, we will not share the data.

REFERENCES:
- [Background] Anderson, N., & West, M. A. (1996). The team climate inventory: Development of the TCI and its applications in team building for innovativeness. European Journal of Work and Organizational Psychology, 5(1), 5366
- [Background] Campion, M. A., Medsker, G. J., & Higgs, A. C. (1993). Relations between work group characteristics and effectiveness: Implications for designing effective work groups. Personnel Psychology, 46(4), 823-847.
- [Background] Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi, D. W., Oishi, S., & Biswas-Diener, R. (2010). New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social Indicators Research, 97, 143-156.
- [Background] Grant AM. Does intrinsic motivation fuel the prosocial fire? Motivational synergy in predicting persistence, performance, and productivity. J Appl Psychol. 2008 Jan;93(1):48-58. doi: 10.1037/0021-9010.93.1.48. PMID 18211134
- [Background] Hadzibajramovic E, Schaufeli W, De Witte H. The ultra-short version of the Burnout Assessment Tool (BAT4)-development, validation, and measurement invariance across countries, age and gender. PLoS One. 2024 Feb 23;19(2):e0297843. doi: 10.1371/journal.pone.0297843. eCollection 2024. PMID 38394265
- [Background] Luthans, F., & Youssef-Morgan, C. M. (2017). Psychological capital: An evidence-based positive approach. Annual Review of Organizational Psychology and Organizational Behavior, 4(1), 339-366.
- [Background] Perugini, M., Gallucci, M., Presaghi, F., & Ercolani, A. P. (2003). The personal norm of reciprocity. European Journal of Personality, 17(4), 251-283.
- [Background] Schaufeli, W. B., Shimazu, A., Hakanen, J., Salanova, M., & De Witte, H. (2017). An ultra-short measure for work engagement. European Journal of Psychological Assessment.
- [Background] Viragos, Anna (2018) Investigating job crafting from a prosocial perspective. PhD thesis, University of Leeds. https://etheses.whiterose.ac.uk/id/eprint/23965/
- See also: This webpage provides general information on the KEEPCARING project. The study registered here is part of this project. — https://keepcaring.eu/

DOCUMENTS (1):
  • Study Protocol (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT06853561/Prot_000.pdf